CLINICAL TRIAL: NCT04409106
Title: The Reliability and Validity of the Turkish Version of the Parental Smartphone Use Management Scale (PSUMS)
Brief Title: The Turkish Version of the Parental Smartphone Use Management Scale (PSUMS)
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ebru Kaya Mutlu, PT, PT, PhD, Assoc Prof., Istanbul University - Cerrahpasa
Other Study IDs: 2020/5
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Addiction Psychological; Addiction; Adolescent
Keywords: Smartphone use; Parental management; Scale validation; Smartphone addiction
MeSH Terms: conditions — Behavior, Addictive; Internet Addiction Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Parental Smartphone Use Management Scale (PSUMS) was originally developed in English language to parents to educate adolescents and communicate with them about online behavior and safety, as well as to conduct plans to manage adolescents' internet and smartphone use. The purpose of this study was to translate and cross-culturally adapt the PSUMS.

DETAILED DESCRIPTION:
Parental Smartphone Use Management Scale (PSUMS) was originally developed in English language to parents to educate adolescents and communicate with them about online behavior and safety, as well as to conduct plans to manage adolescents' internet and smartphone use. The purpose of this study was to translate and cross-culturally adapt the PSUMS. The study will include adults who have been using smartphones for at least the past month and have children aged 11-18. For cross-cultural adaptation, two bi-lingual translators used the back-translation procedure. Within a 5-to-7 day period after first assessment, the participants completed the Turkish version of the Parental Smartphone Use Management Scale (PSUMS) to evaluate test-retest reliability. Cronbach's alpha (α) was used to assess internal consistency. The correlations with the Turkish version of The Smart Phone Addiction Scale-Short Form for Adolescent and the Turkish version of PedsQL in Adolescents 13-18 years old will determine to check the validity.

ELIGIBILITY:
Inclusion Criteria:

* Working at Istanbul University-Cerrahpaşa Faculty of Health Sciences
* Having children using smart phones for at least the last one month
* Having children between aged 11 and 18 years.
* Being a volunteer to participate

Exclusion Criteria:

* Having any serious vision problems or cognitive impairment
* Having disabilities in understanding, speaking and reading Turkish

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The sample will consist of parents who work at Istanbul University-Cerrahpaşa Faculty of Health Sciences and voluntarily agree to participate in the study with children between aged 11 and 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Parental Smartphone Use Management Scale (PSUMS) | Baseline (First assessment)
  Prior to developing the PSUMS, an item pool was established by conducting a literature review and a focus group. The item pool contained 18 items. A 7-point Likert scale was used to rate the level of agreement with items, ranging from 0 (no efficacy at all) to 6 (very strong efficacy).

SECONDARY OUTCOMES:
Parental Smartphone Use Management Scale (PSUMS) | Within a 5-to-7-day period after the first assessment (Second assessment)
  Prior to developing the PSUMS, an item pool was established by conducting a literature review and a focus group. The item pool contained 18 items. A 7-point Likert scale was used to rate the level of agreement with items, ranging from 0 (no efficacy at all) to 6 (very strong efficacy).
Smartphone Addiction Scale -Short form for adolescent Version (SAS-SF) | Baseline (First assessment)
  Smartphone Addiction Scale -Short form for adolescent Version (SAS-SF) is a self-report scale with 10 items rated on a 6-point Likert scale (1= largely untrue, 6= largely true). Higher scores from the scale indicate higher level of the smartphone addiction. . The validity and reliability study of the questionnaire was done in Turkish.
PedsQL in Adolescents | Baseline (First assessment)
  It is a general quality of life scale that evaluates the physical and psychosocial lives of children between the ages of 11-18. The scale prepared for the 13-18 age group has a parent and child form. The parent form is filled out by the caregiver and the adolescent form by the child included in the study separately and simultaneously. The most important features are that "PedsQL in adolescents" is short, it can be filled in about 5-10 minutes, and it is easy to apply and score by the researcher.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru KAYA MUTLU, PhD, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University- Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hsieh YP, Yen CF, Chou WJ. Development and Validation of the Parental Smartphone Use Management Scale (PSUMS): Parents' Perceived Self-Efficacy with Adolescents with Attention Deficit Hyperactivity Disorder. Int J Environ Res Public Health. 2019 Apr 21;16(8):1423. doi: 10.3390/ijerph16081423. PMID 31010068